CLINICAL TRIAL: NCT03671928
Title: Study of Circulating Glicentin Levels in Patients With Intestinal Ischemia
Brief Title: Study of Circulating Levels of Glicentin
Acronym: GLICENTINEDIGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-AOI-12
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Ischemia Bowel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bowel ischemia (Other)
  Interventions: Other: additional blood tube
- non-digestive abdominal pain (Other)
  Interventions: Other: additional blood tube; Other: additional blood sample

INTERVENTIONS:
Other: additional blood tube — sampling of an additional tube at the usual blood test to determine the glicentin level
Other: additional blood sample — for le group control, another blood sample is taken outside the usual care.
  Arms: non-digestive abdominal pain

SUMMARY:
Hormones derived from proglucagon represent a family of peptides produced by the alpha cells of the pancreas and by the intestinal L cells. In the pancreas, the maturation of proglucagon mainly leads to the synthesis of glucagon, while in the intestine, the cleavage of proglucagon allows the synthesis of different peptides including glicentine, oxyntomodulin, Glucagon Like Peptide-1 (GLP-1) and Glucagon Like Peptide-2 (GLP-2).

Glicentin is produced by L cells throughout the digestive tract, from the small intestine to the rectum, with a majority secretion in the colon. Studies in humans and animals have shown its role in the intestinal mucosa. It has a stimulating effect on the proliferation of the intestinal mucosa as well as an effect on smooth muscle cells and regulates trophicity and intestinal motility. Its circulating rate could be modified in case of intestinal ischemia. Mesenteric ischemia is a major diagnostic problem with high morbidity and mortality, particularly in the event of delayed treatment.

The sensitivity and specificity of current markers are low. The identification of new biomarkers of the disease would improve the diagnosis and management of patients with the disease.

The objective of the project is to determine a difference in circulating glicentin levels in patients with intestinal ischemia versus a control group.

On this prospective monocentric study, 40 patients with digestive ischemia will be included in the Emergency Department of the University Hospital of Nice. A control group of 40 patients with abdominal pain will be formed. The circulating glicentin levels will be measured on serum by Elisa technique at the Biochemistry Laboratory of the University Hospital of Nice, work that has been published in 3 scientific journals allowing us to develop and validate the technique.The staff will determine whether patients with digestive ischemia have impaired serum glicentin levels.

The evaluation of the interest of new biological markers of mesenteric ischemia such as glicentine would constitute a definite diagnostic advance. This project could eventually offer new diagnostic and/or therapeutic perspectives in the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* For patients with intestinal ischemia
* The combination of abdominal pain, altered general condition with abdominal defence and venous or arterial hyperlactatemia will be signs suggestive of a diagnosis of digestive ischemia.
* Patients suspected of digestive ischemia with the following comorbidities may be included as clinical suspicion and excluded post-operatively: emboligenic heart disease, arteriopathy, aortic and/or digestive atheromatosis.
* Patients with suspected digestive ischemia and functional scanning ileus.
* Patients with intestinal ischemia proven by CT scan with contrast injection: arterial abnormality such as dissection of an artery for digestive use, thrombosis or embolism of an artery for digestive use; intestinal or colonic thickening suggestive of reversible ischemic suffering of the digestive tract; parietal pneumatosis; gastrointestinal parietal enhancement abnormality (hypo-density ranges or total absence of enhancement).

The following pathologies will be taken into account: mesenteric ischemia by embolism or thrombosis.

* Age over 18 years old
* Able to understand the study
* Affiliation to a social security system
* Signing of an informed consent
* Accept participation in the study (collection of a Non-Opposition)

For the control group

* Age over 18 years old
* Able to understand the study
* Affiliation to a social security system
* Signing of an informed consent
* No personal history of colorectal cancer and obesity
* Admission to the Emergency Department of the University Hospital of Nice for abdominal pain with EVA > 3/10 of non-intestinal origin: nephritic colic, hepatobiliary pathology, gynaecological disease, etc.
* Abdominal CT excluding digestive tract pathology
* Accept participation in the study

Exclusion Criteria:

* History of bariatric or digestive surgery (stomach, small intestine, colon or rectum)
* History of chronic inflammatory bowel disease
* Obese patients (BMI> 30kg/m2)
* History of type 1 diabetes or insulin treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
difference of at least 20% of the serum glicentin dosage in the "intestinal ischemia" group versus the "control" volunteers. | 24 months
  glicentine dosage

CONTACTS AND LOCATIONS:
Locations (1):
- University Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No